CLINICAL TRIAL: NCT02276690
Title: Medical Economic Analysis of the Interest of Hepcidin Quantitation by Quantitative Mass Spectrometry for the Diagnosis of Iron Deficiency in Anemic Critically Ill Patients
Brief Title: Hepcidine and Iron Deficiency in Critically Ill Patients
Acronym: HEPCIDANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 9190
Record Dates: First submitted 2014-10-16; First posted 2014-10-28 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-11

CONDITIONS: Anemia; Critical Illness; Hospitalized for 5 Days or More
Keywords: iron deficiency; dosage of hepcidin; usual biomarker (ferritin and transferrin saturation); mass spectrometry; immuno-detection; anaemia in intensive care unit
MeSH Terms: conditions — Anemia; Critical Illness; Iron Deficiencies | interventions — Hepcidins; Ferritins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dosage of hepcidin (Experimental): In order to assess iron deficiency, patients randomized in this arm will have dosage of hepcidin by mass spectrometry
  Interventions: Biological: hepcidin
- Usual biomarker dosage (Active Comparator): In order to assess iron deficiency, patients randomized in this arm will have usual biomarker dosages (ferritin and transferrin saturation)
  Interventions: Biological: ferritin and transferrin saturation

INTERVENTIONS:
Biological: hepcidin — In order to assess iron deficiency by innovative method (dosage of Hepcidin), an additional collection of blood will be done at day 0 (and weekly until Intensive Care Unit discharge) and at Day 15 after Intensive Care Unit discharge.
  Treatement of Iron deficiency anaemia and anaemia of chronic disease using intravenous iron (± erythropoietin) will be encouraged (or not) according to hepcidin levels
  Arms: Dosage of hepcidin
Biological: ferritin and transferrin saturation — In order to assess iron deficiency by using usual biomarkers (ferritin and transferrin saturation), collection of blood will be done at day 0 (and weekly until Intensive Care Unit discharge) and at Day 15 after Intensive Care Unit discharge.
  Treatement of Iron deficiency anaemia and anaemia of chronic disease using intravenous iron (± erythropoietin) will be encouraged (or not) according to ferritin levels.
  Arms: Usual biomarker dosage

SUMMARY:
Anaemia is very frequent among critically ill patients, concerning more than 60 % of them at admission and more than 80% at intensive care unit discharge. Iron deficiency is also frequent at admission, with prevalence around 25 to 40%. During their stay in Intensive Care Unit, critically ill patients are exposed to repeated blood samples and to other blood losses (daily blood loss has been evaluated to be as high as 128 ml/day in median), this leads to direct iron loss. Prevalence of iron deficiency may thus be very important at Intensive Care Unit discharge. However, iron deficiency diagnosis is complicated in these patients, since inflammation induces an increase in plasma ferritin levels and a decrease in transferrin saturation, the two usual markers of iron deficiency. As a consequence, iron deficiency is usely under-diagnosed in these patients. Treatment of iron deficiency may be indicated to correct anaemia but also to improve patients fatigue and muscular weakness. The characterization of iron metabolism regulation by the hormone hepcidin opened new ways for the understanding and the follow-up of these complex clinical situations (combining inflammation and iron deficiency). Indeed, iron deficiency is associated with a decrease in hepcidin synthesis, while iron overload induces hepcidin synthesis. Furthermore, low hepcidin levels are required to mobilize iron from stores. Hepcidin has thus be proposed as a marker of iron deficiency in critically ill patients. To date, standard immunological methods of hepcidin quantitation are only proposed in the reasearch setting and could not be proposed in the clinical setting because it is too expensive. New approaches for hepcidin quantification, based on mass spectrometry are proposed and may be routinely implemented. We make the hypothesis that treating iron deficiency in critically ill anemic patients, diagnosed by hepcidin quantification, may improve the post-Intensive Care Unit rehabilitation, and may thus reduce post-Intensive Care Unit cost linked to hospital stay and anaemia treatment.

The aim of this study is to evaluate the medical economic interest of a new diagnostic method for iron deficiency, based on a quantitative dosage of hepcidin by mass spectrometry in critically ill anaemic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized man/woman in reanimation unit for at least 5 days.
2. Age ≥ 18 years old.
3. Patient having an anaemia such as defined by the WHO (World Health Organization) (for man: Hemoglobin < 13 g/dl, for woman: Hemoglobin < 12 g/dl).
4. Signed inform consent by the patient or a close person.
5. Subject affiliated to a national health insurance

Exclusion Criteria:

1. Known iron metabolism pathology (such as primitive or secondary hemochromatosis, …).
2. Chronic anaemia (Hemoglobin ≤ 10 g/dl for more than 3 months).
3. Current chemotherapy.
4. Patient having an organ transplant
5. Expected survival < 28 days post Intensive Care Unit discharge.
6. Pregnancy
7. Patient deprived of freedom, by judicial or administrative order.
8. Major protected by the law.
9. Contra-indication to the injectable iron treatment (allergy to ferric carboxymaltose, infection derivates (bacteriamy < 48 hours) untreated).
10. Non speaking French patient, or patient unable to answer a questionnaire because of any neurologic disorder (stroke, brain trauma….).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Hospital cost | from Intensive Care Unit discharge to 90 days after (D90)

SECONDARY OUTCOMES:
Lenght of hospital stay post-Intensive Care Unit | until day 90 after Intensive Care Unit discharge
Haemoglobin levels | 15 days post-Intensive Care Unit discharge
Iron deficiency prevalence | at Day 15 after Intensive Care Unit discharge
Fatigue | 30 days after Intensive Care Unit discharge
  Fatigue will be assessed by the MFI-20 questionnaire
Proportion of patient alive | at Day 90 after Intensive Care Unit discharge
Proportion of patient at home | at Day 90 after Intensive Care Unit discharge
Comparison between mass spectrometry and immuno-detection methods for hepcidin quantification (ancillary study) | from inclusion to Day15 after Intensive Care Unit discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sigismond SL LASOCKI, PU-PH, Study Director — Department of Anesthesiology & Critical Care, Angers University Hospital, France; Sylvain SL LEHMANN, PU-PH, Study Chair — Biochemistry and clinical proteomic laboratory, IRMB, St Eloi University Hospital
Locations (1):
- Department of Anesthesiology & Critical Care, Angers University Hospital, 4 rue larrey, Angers, France

REFERENCES:
- [Background] Lasocki S, Puy H, Mercier G, Lehmann S; Hepcidane study group. Impact of iron deficiency diagnosis using hepcidin mass spectrometry dosage methods on hospital stay and costs after a prolonged ICU stay: Study protocol for a multicentre, randomised, single-blinded medico-economic trial. Anaesth Crit Care Pain Med. 2017 Dec;36(6):391-396. doi: 10.1016/j.accpm.2017.04.009. Epub 2017 Sep 14. PMID 28919067
- [Derived] Lasocki S, Asfar P, Jaber S, Ferrandiere M, Kerforne T, Asehnoune K, Montravers P, Seguin P, Peoc'h K, Gergaud S, Nagot N, Lefebvre T, Lehmann S; Hepcidane study group. Impact of treating iron deficiency, diagnosed according to hepcidin quantification, on outcomes after a prolonged ICU stay compared to standard care: a multicenter, randomized, single-blinded trial. Crit Care. 2021 Feb 15;25(1):62. doi: 10.1186/s13054-020-03430-3. PMID 33588893